CLINICAL TRIAL: NCT06114108
Title: Phase III Randomized Controlled Trial Comparing Maintenance Systemic Therapy Alone With Systemic Therapy Plus Local Ablative Treatment for Patients With Advanced Stage IV Non-small Cell Lung Cancer
Brief Title: Trial Comparing Systemic Therapy Alone and With Local Ablative Treatment for Stage IV NSCL Cancer Patients
Acronym: salVage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: salVage
Record Dates: First submitted 2023-09-22; First posted 2023-11-02 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Stage IV
Keywords: Non-small cell lung cancer (NSCLC); Local consolidative treatment (LAT); patient-reported outcome measures (PROMs)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective, open label, randomized, controlled, multicenter interventional clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Local consolidative treatment (LAT) & Systemic Therapy (Experimental): All patients undergo standard of care (SoC) first-line systemic therapy according to the results of the molecular analysis obtained from the diagnostic biopsy, as per standard of the respective center.
  Patients will undergo additional complete surgical resection of the primary tumor with mediastinal lymph node sampling or radical radiotherapy (preferred stereotactic body radiotherapy (SBRT) to the primary tumor. Surgery and/or SBRT to the metastases will be performed before or after the treatment of the primary tumor according to the clinical need. Thereafter, the treatment will be followed by systemic anticancer treatment as SoC.
  Interventions: Other: Systemic therapy alone or in combination with LAT (surgery and/or radiotherapy); Other: Surgery; Radiation: Radiotherapy
- Control group: Systemic Therapy (Active Comparator): Patients of the control group will receive systemic anticancer treatment alone chemotherapy, chemo-immunotherapy, immunotherapy alone, or targeted treatment).
  Interventions: Other: Systemic therapy alone or in combination with LAT (surgery and/or radiotherapy); Radiation: Radiotherapy

INTERVENTIONS:
Other: Systemic therapy alone or in combination with LAT (surgery and/or radiotherapy) — The choice of LAT intervention for the primary tumor and all metastases (surgery or SBRT) and the sequence of the treatment (primary tumor vs metastases) will be decided at the local MDT according to the medical need and patient counseling during interdisciplinary clinic visits.
  Other Names: Systemic therapy
Other: Surgery — Surgery
  Arms: Intervention group: Local consolidative treatment (LAT) & Systemic Therapy
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
Unfortunately, most patients are already at a very advanced stage when they are diagnosed with lung cancer, i.e. the cancer has already spread outside the lungs forming metastases. The current standard of care therapy at this advanced stage of lung cancer includes systemic anti-cancer therapy such as chemotherapy, immunotherapy to boost the body's immune response, or targeted therapy that directly hinders tumor growth. In this study, the aim is to find out whether it is better if, after a good response to the standard therapy, the remains of main tumor and the metastases are additionally treated by surgery and/or radiation.

DETAILED DESCRIPTION:
In this study, the aim is to find out whether, after a good response to standard therapy, it is better if the main tumor and metastases are additionally removed by surgery and/or radiation. This intervention is referred to as local ablative therapy (LAT). There is evidence to suggest that this additional intervention may prolong the average time to possible cancer recurrence (PFS: Progression-free survival) or lead to longer survival on average. Therefore, the question is to know if these treatments prolong life, and if so, by how much and with what implications. Currently, patients who respond to initial standard therapy are not routinely offered LAT. If the results of this study are positive, it will lead to a fundamental change in the current standard of practice.

The benefit of a therapy is not solely determined by the extension of PFS or overall survival but also heavily influenced by how the therapy impacts patient's quality of life. Medication side effects, pain, fatigue, nausea or extended hospital stays can significantly diminish the perceived positive effects of a treatment from the patient's viewpoint, even if it appears favorable from a medical standpoint. Therefore, the assessment of quality of life through patient-reported outcome measures (PROMs) is a central aspect of this study.

This study will enroll 128 patients from different Swiss hospitals, randomly assigning them to either the intervention group (LAT) or a control group (standard therapy). The study is expected to span approximately two years for each patient.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all of the following inclusion criteria at screening may be enrolled in the trial.

* The inclusion criteria are irrespective from the tumor burden at the time of primary diagnosis before initiation of first line systemic therapy. Neurosurgical diagnostic resection of one single CNS metastasis or laparoscopic resection of one adrenal metastasis before trial inclusion is allowed.
* Adults (18 years or older)
* Tissue confirmed, pre-treatment clinical stage IV NSCLC
* ECOG performance status ≤ 1
* Patients responding after 3 cycles (4th bridging cycle up until randomization is allowed) or 3 months of first line SoC systemic therapy with PR or SD in restaging imaging, and presenting with (induced) oligometastatic or oligopersistent NSCLC defined as a maximum of 5 residual extracranial, distant metastases
* Patients may have up to 5 cranial metastases in addition to the oligoresidual extracranial metastases as long as they are amenable for radiotherapy or surgery.
* The primary tumor and all oligopersistent metastases must be amenable for radical LAT (surgery or radiotherapy)
* Patients of reproductive age agree to use double contraception during the study
* Patient is able to understand trial procedures and is able/willing to adhere to trial procedures as confirmed by signature

Exclusion Criteria:

The presence of any one of the following exclusion criteria at screening will lead to exclusion of the participant:

* Serious concomitant disorder that would compromise patient safety during LAT
* Unresolved complications from initial systemic anticancer treatment, higher than CTCAE grade 2
* Metastatic locations such as malignant ascites, malignant pleural or malignant pericardial effusion, diffuse lymphangiosis of skin or lung, diffuse bone marrow metastasis, abdominal masses/abdominal organomegaly, identified by physical exam that is not measurable by reproducible imaging techniques, leptomeningeal carcinomatosis
* Women who are pregnant or breast feeding
* Patient is currently involved in another trial if either: interventional trial that aims to improve survival, not permitted by other trial, would result in too much patient burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) l in the Local Ablative Therapy (LAT) arm is superior to Standard of Care (SoC) | up to 24 months after randomization
  Progression free survival (PFS) will be assessed by regular clinical examinations of the patients and based on imaging modalities such as (PET)-CT scans and brain MRIs.
Quality of life (QoL) in the LAT arm is non-inferior to the control arm as measured with the European Quality of Life 5 Dimensions 3 Level (EQ-5D-5L) questionnaire-based score at 6 months after randomization | 6 months after randomization
  To show that QoL in the LAT arm is non-inferior to the control arm, mobility the European Quality of Life 5 Dimensions 3 Level (EQ-5D-5L) questionnaire will be used. The questionnaire uses an 1 (no problem) to 5 (extreme problems) scale.

SECONDARY OUTCOMES:
Patients undergoing LAT maintain Quality of Life (QoL) | up to 24 months after randomization
  Patients undergoing LAT maintain Quality of Life (QoL) as measured by using the EQ-5D-5L on different time points of the trial.
To assess safety and tolerability of the LAT strategy as compared to standard of care | from randomization until 30 days after last intervention
  Safety to study interventions will be evaluated by measuring counts of serious adverse events from randomization until 30 days after last intervention or progression, whichever occurs first. Serious adverse events will be evaluated based on CTCAE v5.0.from randomization up until 30 days after last intervention.
To compare quality-adjusted life years | up to 24 months after randomization
  Quality-adjusted life years will be calculated based on the EQ-5D-5L scores and compared between treatment groups, as accrued during the trial observation period across all time points
To evaluate the economic impact of the LAT approach | from signing informed consent until 24 months after randomization
  The economic impact of the LAT approach will be calculated based on the costs of the LAT intervention and on the costs of healthcare utilization outside of the hospital. For the calculation of healthcare utilization costs, patients will be asked on scheduled visits about the healthcare services they have been using outside of the hospital.
To assess the response of primary tumor and metastases to systemic treatment alone and in combination with LAT (according to (i)RECIST criteria) | from intervention until 24 month after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Schmitt-Opitz, Prof, Study Director — Universitätsspital Zürich
Locations (7):
- Switzerland (7):
  - Kantonspital Aarau, Aarau
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Hôpital Fribourgeois - Hôpital Cantonal, Fribourg
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No